CLINICAL TRIAL: NCT00768716
Title: Effect of Race/Ethnicity and Genes on Acetaminophen Pharmacokinetics
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 8600; R01GM061834 (NIH); R01GM102130 (NIH)
Record Dates: First submitted 2008-10-07; First posted 2008-10-08 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2019-05-23 (Actual); Status verified 2019-05

CONDITIONS: Pain; Fever; Hepatotoxicity
MeSH Terms: conditions — Pain; Fever | interventions — Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- White subjects (Experimental): 2 x 500 mg acetaminophen by mouth once
  Interventions: Drug: Acetaminophen
- Black subjects (Experimental): 2 x 500 mg acetaminophen by mouth once
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Acetaminophen — 2 x 500 mg by mouth once
  Other Names: Tylenol

SUMMARY:
Although acetaminophen is the most commonly used nonprescription drug in the USA, little is known regarding the influence of genes and race/ethnicity on acetaminophen disposition. The investigators long-term goal is to understand the causes of differences in acetaminophen disposition between people that are the result of genetic variation and ethnicity and may predispose individuals to a higher risk of acetaminophen hepatotoxicity. The aim of this particular study is to measure the rate of elimination of acetaminophen via the 3 main pathways (glucuronidation, sulfation and oxidation) in self-identified White-Americans (n=100) and African-Americans (n=100). These rates will then be correlated with selected genetic polymorphisms in genes encoding enzymes involved in acetaminophen metabolism. Two main hypotheses will be tested: 1. African-Americans eliminate acetaminophen more rapidly by glucuronidation than do White-Americans. 2. Elimination via glucuronidation, sulfation, and oxidation in subjects will be significantly correlated with the presence of polymorphisms in the UGT1A6, SULT1A1, and CYP2E1 genes, respectively.

ELIGIBILITY:
Inclusion Criteria:

* self-declared white/Caucasian
* self-declared African-American
* active
* ambulatory
* no evidence of medical disease

Exclusion Criteria:

* alcohol use of 3 or more drinks per day
* HIV or hepatitis (B or C) infection
* isoniazid
* disulfiram
* phenobarbital
* phenytoin
* carbamazepine
* rifampicin
* valproic acid
* probenecid
* St. John's Wort

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 95 (Actual)
Dates: Start 2008-12 (Actual); Primary Completion 2012-06 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael H Court, BVSc, PhD, Principal Investigator — Tufts University
Locations (1):
- Tufts Clinical Pharmacology Study Unit, Boston, Massachusetts, United States

REFERENCES:
- [Background] Krishnaswamy S, Hao Q, Al-Rohaimi A, Hesse LM, von Moltke LL, Greenblatt DJ, Court MH. UDP glucuronosyltransferase (UGT) 1A6 pharmacogenetics: I. Identification of polymorphisms in the 5'-regulatory and exon 1 regions, and association with human liver UGT1A6 gene expression and glucuronidation. J Pharmacol Exp Ther. 2005 Jun;313(3):1331-9. doi: 10.1124/jpet.104.081950. Epub 2005 Mar 10. PMID 15761114
- [Background] Krishnaswamy S, Hao Q, Al-Rohaimi A, Hesse LM, von Moltke LL, Greenblatt DJ, Court MH. UDP glucuronosyltransferase (UGT) 1A6 pharmacogenetics: II. Functional impact of the three most common nonsynonymous UGT1A6 polymorphisms (S7A, T181A, and R184S). J Pharmacol Exp Ther. 2005 Jun;313(3):1340-6. doi: 10.1124/jpet.104.081968. Epub 2005 Mar 10. PMID 15761113
- [Background] Court MH, Duan SX, von Moltke LL, Greenblatt DJ, Patten CJ, Miners JO, Mackenzie PI. Interindividual variability in acetaminophen glucuronidation by human liver microsomes: identification of relevant acetaminophen UDP-glucuronosyltransferase isoforms. J Pharmacol Exp Ther. 2001 Dec;299(3):998-1006. PMID 11714888
- [Background] Volak LP, Hanley MJ, Masse G, Hazarika S, Harmatz JS, Badmaev V, Majeed M, Greenblatt DJ, Court MH. Effect of a herbal extract containing curcumin and piperine on midazolam, flurbiprofen and paracetamol (acetaminophen) pharmacokinetics in healthy volunteers. Br J Clin Pharmacol. 2013 Feb;75(2):450-62. doi: 10.1111/j.1365-2125.2012.04364.x. PMID 22725836
- [Background] Court MH, Freytsis M, Wang X, Peter I, Guillemette C, Hazarika S, Duan SX, Greenblatt DJ, Lee WM; Acute Liver Failure Study Group. The UDP-glucuronosyltransferase (UGT) 1A polymorphism c.2042C>G (rs8330) is associated with increased human liver acetaminophen glucuronidation, increased UGT1A exon 5a/5b splice variant mRNA ratio, and decreased risk of unintentional acetaminophen-induced acute liver failure. J Pharmacol Exp Ther. 2013 May;345(2):297-307. doi: 10.1124/jpet.112.202010. Epub 2013 Feb 13. PMID 23408116
- [Background] Court MH, Peter I, Hazarika S, Vasiadi M, Greenblatt DJ, Lee WM; Acute Liver Failure Study Group. Candidate gene polymorphisms in patients with acetaminophen-induced acute liver failure. Drug Metab Dispos. 2014 Jan;42(1):28-32. doi: 10.1124/dmd.113.053546. Epub 2013 Oct 8. PMID 24104197
- [Background] Zhao Y, Harmatz JS, Epstein CR, Nakagawa Y, Kurosaki C, Nakamura T, Kadota T, Giesing D, Court MH, Greenblatt DJ. Favipiravir inhibits acetaminophen sulfate formation but minimally affects systemic pharmacokinetics of acetaminophen. Br J Clin Pharmacol. 2015 Nov;80(5):1076-85. doi: 10.1111/bcp.12644. Epub 2015 Jun 8. PMID 25808818
- [Background] Papageorgiou I, Freytsis M, Court MH. Transcriptome association analysis identifies miR-375 as a major determinant of variable acetaminophen glucuronidation by human liver. Biochem Pharmacol. 2016 Oct 1;117:78-87. doi: 10.1016/j.bcp.2016.08.014. Epub 2016 Aug 13. PMID 27531059
- [Background] Papageorgiou I, Court MH. Identification and validation of microRNAs directly regulating the UDP-glucuronosyltransferase 1A subfamily enzymes by a functional genomics approach. Biochem Pharmacol. 2017 Aug 1;137:93-106. doi: 10.1016/j.bcp.2017.04.017. Epub 2017 Apr 19. PMID 28433553
- [Result] Court MH, Zhu Z, Masse G, Duan SX, James LP, Harmatz JS, Greenblatt DJ. Race, Gender, and Genetic Polymorphism Contribute to Variability in Acetaminophen Pharmacokinetics, Metabolism, and Protein-Adduct Concentrations in Healthy African-American and European-American Volunteers. J Pharmacol Exp Ther. 2017 Sep;362(3):431-440. doi: 10.1124/jpet.117.242107. Epub 2017 Jun 29. PMID 28663312

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | White Subjects | Black Subjects
Started | 54 | 41
Completed | 54 | 41
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | White Subjects | Black Subjects | Total
Number analyzed (Participants) | 54 | 41 | 95
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 54 | 41 | 95
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 43
  Male | 34 | 18 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 41 | 41
  White | 54 | 0 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Acetaminophen Plasma Clearance Association With Race/Ethnicity
Description: Plasma total clearance of acetaminophen in plasma measured by HPLC
Time Frame: 2 days
Measure: Median (Inter-Quartile Range); unit: mL/min/kg
Arm/Group | White Subjects | Black Subjects
Number analyzed (Participants) | 54 | 41
mL/min/kg | 5.3 [4.8 to 6.4] | 5.9 [5.1 to 6.9]
Statistical Analysis 1: Comparison: White Subjects vs Black Subjects; Test type: Other; p = 0.52, Wilcoxon (Mann-Whitney)

2. Primary Outcome: Acetaminophen Glucuronidation Partial Clearance Association With Race/Ethnicity
Description: Acetaminophen glucuronidation partial clearance determined from plasma clearance and urinary metabolite excretion
Time Frame: 2 days
Measure: Median (Inter-Quartile Range); unit: mL/min/kg
Arm/Group | White Subjects | Black Subjects
Number analyzed (Participants) | 54 | 41
mL/min/kg | 2.9 [2.3 to 3.8] | 3.3 [2.4 to 4.1]
Statistical Analysis 1: Comparison: White Subjects vs Black Subjects; Test type: Other; p = 0.42, Wilcoxon (Mann-Whitney)

3. Primary Outcome: Acetaminophen Sulfation Partial Clearance Association With Race/Ethnicity
Description: Acetaminophen sulfation partial clearance determined from plasma clearance and urinary metabolite excretion
Time Frame: 2 days
Measure: Median (Inter-Quartile Range); unit: mL/min/kg
Arm/Group | White Subjects | Black Subjects
Number analyzed (Participants) | 54 | 41
mL/min/kg | 1.4 [1.1 to 1.7] | 1.7 [1.3 to 2.2]
Statistical Analysis 1: Comparison: White Subjects vs Black Subjects; Test type: Other; p = 0.06, Wilcoxon (Mann-Whitney)

4. Primary Outcome: Acetaminophen Oxidation Partial Clearance Association With Race/Ethnicity
Description: Acetaminophen oxidation partial clearance determined from plasma clearance and urinary metabolite excretion
Time Frame: 2 days
Measure: Median (Inter-Quartile Range); unit: mL/min/kg
Arm/Group | White Subjects | Black Subjects
Number analyzed (Participants) | 54 | 41
mL/min/kg | 0.9 [0.65 to 1.15] | 0.57 [0.49 to 0.77]

5. Primary Outcome: Acetaminophen Plasma Clearance Association With UGT2B15 Genotype
Description: The association of UGT2B15 genotype with acetaminophen total clearance
Time Frame: 2 days
Measure: Median (Inter-Quartile Range); unit: mL/min/kg
Groups:
- UGT2B15*1/*1; UGT2B15*1/*2; UGT2B15*2/*2: UGT2B15 genotype
Arm/Group | UGT2B15*1/*1 | UGT2B15*1/*2 | UGT2B15*2/*2
Number analyzed (Participants) | 27 | 45 | 22
mL/min/kg | 6.4 [5.4 to 7.7] | 5.5 [4.9 to 6.5] | 4.7 [4.2 to 5.3]
Statistical Analysis 1: Comparison: UGT2B15*1/*1 vs UGT2B15*1/*2 vs UGT2B15*2/*2; Test type: Other; p < 0.0001, ANOVA

6. Primary Outcome: Acetaminophen Glucuronidation Partial Clearance Association With UGT2B15 Genotype
Description: The association of acetaminophen glucuronidation partial clearance with UGT2B15 genotype
Time Frame: 2 days
Measure: Median (Inter-Quartile Range); unit: mL/min/kg
Arm/Group | UGT2B15*1/*1 | UGT2B15*1/*2 | UGT2B15*2/*2
Number analyzed (Participants) | 27 | 43 | 22
mL/min/kg | 3.8 [2.7 to 4.0] | 2.8 [2.2 to 3.9] | 2.1 [1.4 to 2.7]
Statistical Analysis 1: Comparison: UGT2B15*1/*1 vs UGT2B15*1/*2 vs UGT2B15*2/*2; Test type: Other; p < 0.0001, ANOVA

7. Primary Outcome: APAP Plasma Adduct Association With UGT2B15 Genotype
Description: The association of UGT2B15 genotype with APAP plasma adduct concentrations
Time Frame: 2 days
Measure: Median (Inter-Quartile Range); unit: mL/min/kg
Arm/Group | UGT2B15*1/*1 | UGT2B15*1/*2 | UGT2B15*2/*2
Number analyzed (Participants) | 27 | 44 | 21
mL/min/kg | 16 [11 to 23] | 19 [13 to 26] | 27 [21 to 35]
Statistical Analysis 1: Comparison: UGT2B15*1/*1 vs UGT2B15*1/*2 vs UGT2B15*2/*2; Test type: Other; p = 0.003, ANOVA

ADVERSE EVENTS:
Time Frame: 2 days
Arm/Group | White Subjects | Black Subjects
All-Cause Mortality (participants affected / at risk) | 0/54 | 0/41
Serious Adverse Events (participants affected / at risk) | 0/54 | 0/41
Other Adverse Events (participants affected / at risk) | 0/54 | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes